CLINICAL TRIAL: NCT07382271
Title: Evaluation of Safety and Efficacy of Phage Therapy for Drug-resistant Bacterial Infections: An Exploratory, Prospective Single-arm Study
Acronym: Phage Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJT2025V2.0; 20250901 (Other Grant/Funding Number: Jiangsu Jicui Medical Engineering Cross Technology Research Institute Co., Ltd.)
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Urinary Tract Infections; Urinary Tract Infections Caused by Drug-resistant Bacteria
Keywords: Phage Therapy; Drug-resistant bacteria; Urinary tract infection; Personalized phage cocktail
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Phage Cocktail Therapy for Drug-Resistant Urinary Tract Infections (Experimental): This arm enrolls eligible patients with drug-resistant bacterial urinary tract infections (UTIs). The core intervention is personalized phage cocktail therapy, tailored to each patient's isolated drug-resistant pathogen (e.g., carbapenem-resistant Acinetobacter baumannii, Klebsiella pneumoniae, Pseudomonas aeruginosa; vancomycin-resistant Enterococcus; methicillin-resistant Staphylococcus aureus; Stenotrophomonas maltophilia).
  Key Details of the Intervention:
  1. Phage Cocktail Preparation: Target pathogens isolated from patients' urine samples undergo in vitro lytic phage matching via double-layer agar plate assay or liquid killing curve assay. The cocktail is formulated using lytic phages screened from a high-quality phage library (provided by Chuangshiji (Shanghai) Biotechnology Co., Ltd.), following the group standard T/SHPPA 028-2024 (Quality Requirements for Clinical Therapeutic Bacteriophage Preparations). Each batch is purified and packaged in GMP-compliant facilities, with a s
  Interventions: Biological: Personalized Phage Cocktail

INTERVENTIONS:
Biological: Personalized Phage Cocktail — Intravesical perfusion via urinary catheter. 50 mL of diluted phage cocktail (diluted with Ringer's solution if needed) is infused, followed by clamping the catheter for 30 minutes to maximize phage-bacteria contact. Dosing is repeated every 12 hours for 2 or 3 consecutive days (6 total doses).

SUMMARY:
This study is an investigator-initiated, single-center, exploratory clinical trial designed to evaluate the safety and efficacy of phage therapy in patients with urinary tract infections caused by drug-resistant bacteria.

Eligible patients aged 18 to 65 years will receive the phage cocktail intervention according to a predefined dosage regimen, with a treatment course of 2 to 3 days and a follow-up period of 2 to 4 weeks after treatment. The primary outcome measures include the incidence of adverse events during treatment, the pathogen clearance rate, and the improvement of clinical symptoms (e.g., fever, local inflammation).

The purpose of this study is to provide a scientific basis for the subsequent clinical application of this phage cocktail, and to explore a novel therapeutic option for patients with drug-resistant bacterial infections who have shown poor responses to conventional antibiotic therapy. All participants will undergo standardized medical monitoring throughout the trial, and their rights and safety will be fully protected by the Institutional Review Board (IRB) during the entire process.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, single-arm exploratory clinical study conducted at the Department of Infectious Diseases, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School. The study aims to systematically evaluate the safety and efficacy of personalized phage cocktail therapy in patients with urinary tract infections (UTIs) caused by drug-resistant bacteria, addressing the unmet clinical need for alternative treatments amid the global spread of antibiotic resistance.

1. Study Rationale Global mortality associated with drug-resistant bacterial infections reached 4.95 million in 2019, with 1.27 million deaths directly attributed to this cause. Projections indicate this number could rise to 10 million annually by 2050 without effective interventions. The development of new antibiotics lags far behind the emergence of drug-resistant strains, as most newly approved agents are derivatives of existing antibiotics with established resistance mechanisms. Phage therapy, leveraging the natural specificity of bacteriophages to lyse target bacteria without harming human cells or the commensal microbiota, has emerged as a promising alternative. Clinical evidence from over 6,300 global cases and systematic reviews confirms its favorable safety profile (7.5% adverse event rate vs. 14.9% for conventional antibiotics) and efficacy (78.8% clinical improvement rate, 86.7% pathogen clearance rate). This study builds on these findings to validate the clinical applicability of personalized phage therapy for drug-resistant UTIs.
2. Study Design and Scope

   * Study Type: Prospective, single-arm, exploratory study without a control group (justified by ethical considerations and the lack of standardized control protocols for novel phage therapy).
   * Sample Size: 6 eligible patients (determined based on prior clinical data and institutional capacity).
   * Study Period: Each participant undergoes a screening period (≤7 days), a treatment period (2-3 days), and a follow-up period (2-4 weeks), with a total observation duration of up to 5 weeks.
   * Study Site: Department of Infectious Diseases, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Nanjing, China).
3. Eligibility Criteria 3.1 Inclusion Criteria

<!-- -->

1. Aged 18-65 years old.
2. Patients with urinary tract infections caused by drug-resistant bacteria (based on drug susceptibility test results from our hospital or other Grade A tertiary hospitals).
3. The pathogenic bacteria infected by the patient must meet one of the following conditions:

   a) Pathogenic bacteria are resistant to key antibiotics:
   * Acinetobacter baumannii: carbapenem-resistant;

     * Enterobacteriaceae (e.g., Klebsiella pneumoniae, Escherichia coli): carbapenem or cephalosporin-resistant; ③ Pseudomonas aeruginosa: carbapenem-resistant;

       ④ Enterococci: vancomycin-resistant;

       ⑤ Staphylococcus aureus: methicillin or vancomycin-resistant;
       * Stenotrophomonas maltophilia. Referenced to the WHO Bacterial Priority Pathogens List, 2024 b) The pathogenic bacteria are sensitive to key antibiotics in vitro, but treatment with such antibiotics is ineffective or shows insignificant efficacy (the patient's target bacterial infection persists for 7 days or more, and the infection cannot be eradicated despite antibiotic administration during this period).

         c) The use of key antibiotics to which the pathogenic bacteria are sensitive is restricted (e.g., potential organ toxicity caused by the antibiotics, or the patient is allergic to such antibiotics).
4. At least one lytic phage targeting the pathogenic bacteria can be screened out.
5. The patient can tolerate the procedures of intravesical perfusion via urinary catheter, retrograde pyeloperfusion via ureteral catheter, or pyeloperfusion via percutaneous nephrostomy tube, and agrees to receive indwelling or intermittent catheterization during the treatment period.
6. The subject and their family members (or legal guardian) have fully read and understood the relevant information, and signed the informed consent form.

3.2 Exclusion Criteria

1. Bacterial infection controllable with conventional antibiotic therapy.
2. Presence of undrained urinary tract abscess or obstruction.
3. Severe renal impairment (eGFR <30 mL/min/1.73m²).
4. Concurrent organ failure (heart, liver, lung, etc.).
5. Severe autoimmune diseases.
6. No available phages active against the infecting pathogen.
7. Other conditions deemed unsuitable by the investigator.

4. Intervention Details 4.1 Phage Preparation

* Test Product: Personalized phage cocktail provided by Chuangshiji (Shanghai) Biotechnology Co., Ltd., consisting of lytic phages targeting the participant's specific pathogen. The formulation is purified and packaged in GMP-compliant facilities, with a specification of 5 mL/vial and a titer ≥10⁷ PFU/mL.
* Phage Matching: Pathogens isolated from participants are sent to a collaborative laboratory for high-throughput phage screening using double-layer agar plate assay or liquid killing curve assay. The Next Evolution Phage-Typing (NEPT) method is preferred to combine primary and secondary phages, preventing the emergence of phage-resistant bacteria.
* Quality Control: Each batch undergoes sterility testing (48-hour culture on blood agar plates with no bacterial growth) and titer verification using the participant's target pathogen (≥10⁷ PFU/mL, per the group standard T/SHPPA 028-2024).

4.2 Administration

Treatment routes are selected based on infection location:

• Intravesical Perfusion (for lower UTIs): 50 mL of phage cocktail (diluted with Ringer's solution if needed) is infused via urinary catheter. The catheter is clamped for 30 minutes post-administration, then removed or unclamped. Dosing is repeated every 12 hours for 4-6 total doses (2 or 3-day course).

4.3 Concomitant Medications Antibiotics may be administered based on susceptibility testing and clinical judgment. If no susceptible antibiotics are available, the Non-active Antibiotic and Bacteriophage Synergism (NABS) method is used to identify antibiotics with synergistic effects with phages.

5. Outcome Measures 5.1 Safety Outcomes

* Primary Safety Endpoints: Incidence, severity, and causality of adverse events (AEs) and serious adverse events (SAEs) during treatment and follow-up. Key monitored events include:

  o Bacteriolysis-related reactions (e.g., endotoxin release syndrome: fever >39℃, hypotension).
  * Immunogenic reactions (e.g., rash, dyspnea, anaphylaxis).
* Safety Assessments: Vital signs (daily during treatment); laboratory tests (complete blood count, liver/kidney function, CRP, procalcitonin, cytokines) at baseline, Day 1, 3, 5, and 7 post-treatment; and clinical observations for AEs.

5.2 Efficacy Outcomes

* Primary Efficacy Endpoint: Pathogen clearance rate, defined as:

  o Negative urine culture for the target pathogen in two consecutive samples, or

  o ≥10-fold reduction in bacterial load (absolute quantification) or ≥2-grade reduction in semi-quantification (4-quadrant streaking method) if the pathogen persists.
  * Assessments are conducted at baseline and Days 1, 3, 5, 7 post-treatment.
* Secondary Efficacy Endpoint: Clinical symptom resolution rate, evaluated as:

  o Complete resolution: Disappearance of dysuria, frequency, urgency, lumbago, and fever; normal urine routine (leukocytes <5/HPF, nitrite negative); negative urine culture.

  o Partial resolution: Improvement in symptoms with mild residual abnormalities.

  o Assessments are performed at each follow-up visit (Weeks 1, 2, 3, 4 post-treatment).

  6. Safety Monitoring and Ethical Protection
* AE/SAE Management: All AEs are documented, tracked, and graded per CTCAE criteria. SAEs (e.g., death, life-threatening events, hospitalization) are reported to the Institutional Review Board (IRB) within 24 hours.
* Ethical Compliance: The study complies with the Declaration of Helsinki and GCP guidelines. The protocol has been approved by the Medical Ethics Committee of The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School. Participants may withdraw at any time without penalty.
* Data Safety Monitoring: The principal investigator conducts regular reviews of accumulated safety data to assess risk-benefit balance and recommend study continuation or termination if necessary.

  7. Study Timeline
* January 2026 - June 2026: Patient screening, enrollment, treatment, and follow-up.
* July 2026 - August 2026: Data analysis and study report completion.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-65 years old. 2. Patients with urinary tract infections caused by drug-resistant bacteria (based on drug susceptibility test results from our hospital or other Grade A tertiary hospitals).

  3. The pathogenic bacteria infected by the patient must meet one of the following conditions:
  1. Pathogenic bacteria are resistant to key antibiotics:

     ① Acinetobacter baumannii: carbapenem-resistant;
     * Enterobacteriaceae (e.g., Klebsiella pneumoniae, Escherichia coli): carbapenem or cephalosporin-resistant;

       * Pseudomonas aeruginosa: carbapenem-resistant;

         * Enterococci: vancomycin-resistant; ⑤ Staphylococcus aureus: methicillin or vancomycin-resistant; ⑥ Stenotrophomonas maltophilia. Referenced to the WHO Bacterial Priority Pathogens List, 2024
  2. The pathogenic bacteria are sensitive to key antibiotics in vitro, but treatment with such antibiotics is ineffective or shows insignificant efficacy (the patient's target bacterial infection persists for 7 days or more, and the infection cannot be eradicated despite antibiotic administration during this period).
  3. The use of key antibiotics to which the pathogenic bacteria are sensitive is restricted (e.g., potential organ toxicity caused by the antibiotics, or the patient is allergic to such antibiotics).

     4. At least one lytic phage targeting the pathogenic bacteria can be screened out.

     5. The patient can tolerate the procedures of intravesical perfusion via urinary catheter, retrograde pyeloperfusion via ureteral catheter, or pyeloperfusion via percutaneous nephrostomy tube, and agrees to receive indwelling or intermittent catheterization during the treatment period.

     6. The subject and their family members (or legal guardian) have fully read and understood the relevant information, and signed the informed consent form.

     Exclusion Criteria:
* 1. Bacterial infection controllable with conventional antibiotic therapy. 2. Presence of undrained urinary tract abscess or obstruction. 3. Severe renal impairment (eGFR <30 mL/min/1.73m²). 4. Concurrent organ failure (heart, liver, lung, etc.). 5. Severe autoimmune diseases. 6. No available phages active against the infecting pathogen. 7. Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pathogen Clearance Rate | Baseline (pre-treatment); Days 1, 3, 5, 7 post-treatment

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected in this trial will be shared after the publication of the primary study results, to support further scientific research on phage therapy for drug-resistant urinary tract infections. The shared data will be de-identified to protect participant privacy (removal of names, identification numbers, contact information, and other personal identifiers).
  The shared dataset will include: baseline demographic data, pathogen identification and drug susceptibility test results, outcome measure data (pathogen clearance rate, clinical symptom resolution rate, adverse event records), and intervention administration records. The study protocol, statistical analysis plan, and informed consent form will also be made publicly available.
  Eligible researchers may request access to the IPD by submitting a research proposal to the study's data access committee. The proposal should specify the research objectives, analysis methods, and expected outputs. Data will be
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code